CLINICAL TRIAL: NCT01525823
Title: Effects of Metformin on Glucose Homeostasis Following Administration of BMS-754807 in Healthy Volunteer Subjects
Brief Title: Assessment of Blood Glucose Changes in Healthy Volunteers After BMS-754807 Alone or BMS-754807 With Metformin
Acronym: NHV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CA191-015
Record Dates: First submitted 2012-01-18; First posted 2012-02-03 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — BMS 754807; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BMS-754807 + Metformin (Experimental)
  Interventions: Drug: BMS-754807 (IGR-IR/IR Inhibitor); Drug: Metformin

INTERVENTIONS:
Drug: BMS-754807 (IGR-IR/IR Inhibitor) — Tablets, Oral, 100mg, Once daily, Days 1 - 5 and 15 - 17
Drug: Metformin — Tablets, Oral, (1000mg on Days 3 - 9) and (2000mg on Days 10 - 17), Once daily

SUMMARY:
The purpose of this study is to assess the effects of Metformin administered over two weeks on the peak plasma glucose concentrations following administration of BMS-754807.

DETAILED DESCRIPTION:
Primary Purpose: Other - Protocol designed to evaluate pharmacodynamics following administration of two compounds

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects ages 18 to 55 determined with no clinically significant deviation from normal medical history, physical examination, electrocardiograms (ECGs), and clinical laboratory
* Women who are not of childbearing potential

Exclusion Criteria:

* Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG or clinical laboratory determinations consistent with a healthy volunteer target population
* History of clinically relevant hypoglycemic events
* History of clinically relevant hyperglycemic events

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2012-02; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Mean difference of the peak plasma glucose concentrations following administration of BMS-754807 alone and following 2 weeks of Metformin administration | On Day 3 and Day 17

SECONDARY OUTCOMES:
Safety endpoints: AEs and marked clinical laboratory abnormalities | Day -21 to Day 47
  Incidence of adverse events (AEs), AEs leading to discontinuation, serious adverse events (SAEs), and deaths occurring up to 30 days after the last dose of study medication and marked abnormalities of laboratory values
Maximum observed plasma concentration (Cmax) of BMS-754807 and M5 | 9 timepoints over 24 hours following Day 1 dose and 12 timepoints over 72 hours for the Day 5 dose
Time of maximum observed plasma concentration (Tmax) of BMS-754807 and M5 | 9 timepoints over 24 hours following Day 1 dose and 12 timepoints over 72 hours for the Day 5 dose
Area under the plasma concentration-time curve from time zero extrapolated to infinite time [AUC(INF)] of BMS-754807 and M5 | 12 timepoints over 72 hours for the Day 5 dose
Area under the plasma concentration-time curve in one dosing interval [AUC(TAU)] of BMS-754807 and M5 | 9 timepoints over 24 hours following Day 1 dose and 12 timepoints over 72 hours for the Day 5 dose
Area under the plasma concentration-time curve from time zero to the last quantifiable plasma concentration [AUC(0-T)] of BMS-754807 and M5 | 9 timepoints over 24 hours following Day 1 dose and 12 timepoints over 72 hours for the Day 5 dose
Plasma half-life (T-HALF) of BMS-754807 and M5 | 12 timepoints over 72 hours for the Day 5 dose
Accumulation index; ratio of AUC(TAU) at steady-state to AUC(TAU) after the first dose (AI) of BMS-754807 and M5 | 9 timepoints over 24 hours following Day 1 dose and 12 timepoints over 72 hours for the Day 5 dose
Mean levels of plasma glucose, serum insulin and c-peptide | Day 3, Day 5 and Day 17

CONTACTS AND LOCATIONS:
Overall Officials: Bristol_Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Melbourne, Victoria, Australia